CLINICAL TRIAL: NCT01413100
Title: A Phase II Multi-center Study of High-Dose Cyclophosphamide and Antithymocyte Globulin Followed by Autologous Hematopoietic Cell Transplantation With Post Transplant Maintenance for the Treatment of Systemic Sclerosis
Brief Title: Scleroderma Treatment With Autologous Transplant (STAT) Study
Acronym: STAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Leona Holmberg, Professor, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2533.00; NCI-2011-01190 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2533; 2533.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG1711052 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2011-08-08; First posted 2011-08-10 (Estimated); Results first posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Systemic Scleroderma
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Antilymphocyte Serum; thymoglobulin; Cyclophosphamide; Filgrastim; Granulocyte Colony-Stimulating Factor; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; plerixafor; ferric pyrophosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (HDIT autologous PBSCT) (Experimental): STEM CELL MOBILIZATION AND PREPARATION: Patients receive filgrastim SC on mobilization days 1-4 followed by apheresis until a target dose of CD34+ cells >= 2.5 x 10^6/kg are collected. Patients difficult to mobilize with filgrastim alone receive cyclophosphamide IV or *plerixafor SC on mobilization days 1-2 and filgrastim SC on mobilization days 5-7.
  HDIT CONDITIONING: Patients receive high-dose cyclophosphamide IV over 1-2 hours on days -5 to -2 and anti-thymocyte globulin IV on days -5, -3, -1, 1, 3, and 5.
  TRANSPLANTATION: Patients undergo autologous PBSCT on day 0.
  MAINTENANCE THERAPY: Beginning 2-3 months after transplant, patients receive mycophenolate mofetil PO BID for 2 years.
  Interventions: Biological: Anti-Thymocyte Globulin; Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Cyclophosphamide; Biological: Filgrastim; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Peripheral Blood Stem Cell Transplantation; Drug: Plerixafor; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Biological: Anti-Thymocyte Globulin — Given IV
  Other Names: Antithymocyte Globulin; Antithymocyte Serum; ATG; ATGAM; ATS; Thymoglobulin
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo autologous PBSCT
  Other Names: Autologous Stem Cell Transplantation
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Biological: Filgrastim — Given SC
  Other Names: Filgrastim XM02; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tbo-filgrastim; Tevagrastim
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mycophenolate Mofetil — Given PO
  Other Names: Cellcept; MMF
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo autologous PBSCT
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplantation
Drug: Plerixafor — Given SC
  Other Names: AMD 3100; JM-3100; Mozobil; SDZ SID 791
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well giving cyclophosphamide and anti-thymocyte globulin together followed by peripheral blood stem cell transplant (PBSCT) and mycophenolate mofetil works in treating patients with systemic scleroderma (SSc). Stem cells are collected from the patient's blood and stored prior to treatment. To store the stem cells patients are given colony-stimulating factors, such as filgrastim (G-CSF) or chemotherapy (cyclophosphamide) to help stem cells move from the bone marrow to the blood so they can be collected and stored. After storage, patients are then given high-dose chemotherapy, cyclophosphamide, and immunosuppression with anti-thymocyte globulin to suppress the immune system to prepare for the transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy and immunosuppression. After the stem cells have "engrafted" and have matured enough to support the immune system at approximately 2-3 months, patients are given a medication called mycophenolate mofetil (MMF) or Myfortic. This medication is given to prevent worsening or reactivation of SSc and is referred to as maintenance therapy.

DETAILED DESCRIPTION:
OUTLINE:

STEM CELL MOBILIZATION AND PREPARATION: Patients receive filgrastim subcutaneously (SC) on mobilization days 1-4 followed by apheresis until a target dose of CD34+ cells >= 2.5 x 10^6/kg are collected. Patients difficult to mobilize with filgrastim alone receive cyclophosphamide intravenously (IV) or *plerixafor subcutaneously (SC) on mobilization days 1-2 and filgrastim SC on mobilization days 5-7.

HDIT CONDITIONING: Patients receive high-dose cyclophosphamide IV over 1-2 hours on days -5 to -2 and anti-thymocyte globulin IV on days -5, -3, -1, 1, 3, and 5.

TRANSPLANTATION: Patients undergo autologous PBSCT on day 0.

MAINTENANCE THERAPY: Beginning 2-3 months after transplant, patients receive mycophenolate mofetil orally (PO) twice daily (BID) for 2 years.

NOTE: *Plerixafor is an alternative to the cyclophosphamide based mobilization.

After completion of study treatment, patients are followed at 1 month, weeks 12 and 26, and then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with SSc as defined by the American College of Rheumatology with diffuse cutaneous disease (except Group 5) at risk of disease progression
* Patients must have failed a prior >= 4-mponth course of either MMF/Myfortic or cyclophosphamide before being eligible for the study (determined at >= 1 week before start of mobilization); "failure" is defined as evidence of disease progression or absence of improvement; the response prior to MMF of cyclophosphamide will be assessed by the participating site study rheumatologist
* Patients must meet eligibility in at least 1 of the following 6 groups:
* GROUP 1:

  * Patients must have 1) both a and b below; and 2) either c, or d

    * a) Diffuse cutaneous scleroderma as defined by skin thickening proximal to the elbows and knees and/or involving the torso in addition to distal extremity involvement; a skin score will be obtained but not used to determine eligibility
    * b) Duration of systemic sclerosis =< 7 years from the onset of first non-Raynaud's symptom; for those patients with disease activity between 5-7 years from the onset of first non-Raynaud's symptom, recent progression or activity of disease must be documented
    * c) Presence of SSc-related pulmonary disease with forced vital capacity (FVC) < 80% or hemoglobin-adjusted diffusing capacity for carbon monoxide (DLCO) < 70% of predicted AND evidence of alveolitis or SSc-related interstitial lung disease by high-resolution chest computed tomography (CT) scan and/or by bronchoalveolar lavage (BAL) (interstitial lung disease may be nonspecific interstitial pneumonia [NSIP] or usual interstitial pneumonia [UIP]; a bronchoalveolar lavage [BAL] should be done to confirm the findings of alveolitis only if the high resolution CT scan [HRCT] fails to show findings typically associated with systemic sclerosis changes [ground glass NSIP, UIP, SSc related interstitial lung disease]); alveolitis by BAL cell count will be defined based on a BAL cell differential count (> 3% neutrophils and/or > 2% eosinophils) from any lavaged lobe
    * d) History of SSc-related renal disease that may not be active at the time of screening; stable serum creatinine must be documented for a minimum of 3 months post-renal crisis at the time of the baseline visit; history of scleroderma hypertensive renal crisis is included in this criterion and is defined as follows:

      * History of new-onset hypertension based on any of the following (measurements must be repeated and confirmed at least 2 hours apart within 3 days of first event-associated observation, with a change from baseline):

        * Systolic blood pressure (SBP) >= 140 mmHg
        * Diastolic blood pressure (DBP) >= 90 mmHg
        * Rise in SBP >= 30 mmHg compared to baseline
        * Rise in DBP >= 20 mmHg compared to baseline
      * AND one of the following 5 laboratory criteria:

        * Increase of >= 50 % above baseline in serum creatinine

          * Proteinuria: >= 2+ by dipstick confirmed by protein:creatinine ratio > 2.5
          * Hematuria: >= 2+ by dipstick or > 10 red blood cell (RBC)s/hematopoietic-promoting factor (HPF) (without menstruation)
          * Thrombocytopenia: < 100,000 platelets/mm^3
          * Hemolysis: by blood smear or increased reticulocyte count
      * The above definition of SSc hypertensive renal crisis is independent of whether concomitant anti-hypertensive medications are used
      * Subjects who present with solely skin and renal disease in the absence of other organ involvement, except classic SSc renal crisis as described above and including non-hypertensive renal crisis, must see a nephrologist to confirm that their renal disease is secondary to only SSc
      * Note: Subjects may be re-screened if they fail to meet inclusion criteria on initial evaluation
* GROUP 2:

  * Progressive pulmonary disease as defined by a decrease in the FVC or DLCO-adjusted by 10 or 15 percent or greater, respectively, from a prior FVC or DLCO-adjusted in the previous 18-month period
  * Patients will have diffuse cutaneous disease and may have both FVC and DLCOcorr >= 70% at screening for the study
  * Patients must also have evidence of alveolitis as defined by abnormal chest computed tomography (CT) or bronchoalveolar lavage (BAL)
* GROUP 3: Diffuse scleroderma with disease duration =< 2 years since development of first sign of skin thickening plus modified Rodnan skin score >= 25 plus either

  * Erythrocyte sedimentation rate (ESR) > 25 mm/1st hour and/or hemoglobin (Hb) < 11 g/dL, not explained by causes other than active scleroderma
  * Lung involvement (either FVC or DLCO < 80% and evidence of interstitial lung disease by CT scan or alveolitis by BAL)
* GROUP 4: Diffuse scleroderma with disease duration =< 2 years and skin score >= 30
* GROUP 5:

  * Limited cutaneous scleroderma and SSc-related pulmonary disease with FVC < 80% or hemoglobin-adjusted DLCO < 70% of predicted
  * AND evidence of alveolitis/interstitial lung disease by high-resolution chest CT scan and/or by BAL (interstitial lung disease may be nonspecific interstitial pneumonia [NSIP] or usual interstitial pneumonia [UIP]; A bronchoalveolar lavage [BAL] should be done to confirm the findings of alveolitis only if the high resolution CT scan [HRCT] fails to show findings typically associated with systemic sclerosis changes [ground glass, NSIP, UIP, SSc related interstitial lung disease])
  * Alveolitis by BAL cell count will be defined based on a BAL cell differential count (> 3% neutrophils and/or > 2% eosinophils) from any lavaged lobe
* GROUP 6: Progressive gastrointestinal disease as defined by all of the following items:

  * Disease duration of scleroderma =< 2 years.
  * Documented severe malabsorption syndrome requiring nutritional support; severe malabsorption syndrome is > 10% weight loss and on total parenteral nutrition (TPN) or enteral feedings
  * High score on distention/ bloating scale (>= 1.60 out of 3.00) on gastrointestinal (GI) questionnaire

Exclusion Criteria:

* Subjects with pulmonary, cardiac, hepatic, or renal impairment that would limit their ability to receive cytoreductive therapy and compromise their survival; this includes, but is not restricted to, subjects with any of the following:
* Pulmonary dysfunction defined as:

  * Severe pulmonary dysfunction with (1) a hemoglobin corrected DLCO < 40% of predicted at the Baseline Screening visit, or (3) FVC < 45% of predicted Baseline Screening visit, or
  * Partial pressure (pO2) < 70 mmHg or pCO2 >= 45 mmHg without supplemental oxygen, or
  * O2 saturation < 92% at rest without supplemental oxygen as measured by forehead pulse oximeter
* Significant pulmonary artery hypertension (PAH) defined as:

  * Peak systolic pulmonary artery pressure > 50 mmHg by resting echocardiogram will require right heart catheterization; if pulmonary artery pressure (PAP) is not evaluable on echocardiogram due to lack of a Tricuspid regurgitant jet, then normal anatomy and function as evidenced by normal right atrium and ventricle size, shape and wall thickness and septum shape must be documented to rule-out PAH; otherwise, right heart catheterization is indicated; prior history of PAH but controlled with medications will not exclude patients from the protocol; PAH is considered controlled with medications if peak systolic pulmonary artery pressure is < 45 mmHg or mean pulmonary artery pressure by right heart catheterization is < 30 mmHg at rest
  * Mean pulmonary artery pressure by right heart catheterization exceeding 30 mmHg at rest; if mean PAP is elevated and pulmonary vascular resistance and transpulmonary gradient are normal then the patient is eligible for the protocol
  * New York Heart Association (NYHA)/World Health Organization Class III or IV
* Cardiac: Uncontrolled clinically significant arrhythmias; clinical evidence of significant congestive heart failure (CHF) (NYHA Class III or IV); left ventricular ejection fraction (LVEF) < 50% by echocardiogram
* History/presence of arrhythmia (even controlled) on chemical anti-arrhythmic(s) must have cardiac consult to ensure the subject could safely proceed with protocol requirements
* Significant renal pathology defined as:

  * Estimated creatinine clearance (CrCl) < 40 mL/min (using Cockcroft-Gault formula based on actual body weight) and serum creatinine > 2.0 mg/dL; OR
  * Active, untreated SSc renal crisis at the time of enrollment; presence of nephrotic range proteinuria (defined as >= 3.5 gms/24 hours, or protein:creatinine ratio >= 3.5), active urinary sediment, urinary RBCs > 25 per HPF, or red cell casts require further investigation by a nephrologist to rule out glomerulonephritis, overlap syndromes, or other causes of renal disease in all subjects; subjects with glomerulonephritis or overlap syndromes will be excluded
* Hepatic: Active hepatitis (alanine aminotransferase [ALT], aspartate aminotransferase [AST], or bilirubin > 2 times the upper limit of normal [ULN]) or evidence of moderate to severe periportal fibrosis by liver biopsy
* Active or clinically significant Gastric Antral Vascular Ectasia (GAVE, "watermelon stomach")
* Unwilling or unable to discontinue disallowed disease-modifying antirheumatic drugs (DMARDs) for treatment of SSc prior to mobilization
* History or presence of a 2nd autoimmune disease requiring immunosuppressive therapy that has substantial risk of immunosuppressive treatment beyond transplant with the following exceptions:

  * History and/or presence of Sjogren's Syndrome is allowed
  * Stable myositis (A history of myositis that is clinically stable as defined by lack of progressive proximal muscle weakness and a stable or decreasing creatine phosphokinase [CPK] < 3 x ULN) is allowed
  * The presence of anti-double stranded (ds)-deoxyribonucleic acid (DNA) without clinical systemic lupus erythematosus in a patient with a diagnosis of otherwise "pure" SSc is allowed
  * Concomitant rheumatoid arthritis without extra-articular disease characteristic of rheumatoid arthritis is allowed
* Active uncontrolled infection that would be a contraindication to safe use of high-dose therapy
* Positive study for Hepatitis B surface antigen or Hepatitis B or C confirmed by polymerase chain reaction (PCR)
* Positive serology for human immunodeficiency virus (HIV)
* Absolute neutrophil count (ANC) < 1500 cells/uL
* Platelets < 100,000 cells/uL
* Hematocrit < 27%
* Hemoglobin < 9.0 g/dL
* Malignancy within the 2 years prior to entry in study, excluding adequately treated squamous cell skin cancer, basal cell carcinoma, and carcinoma in situ; treatment must have been completed (with the exception of hormonal therapy for breast cancer) with cure/remission status verified for at least 2 years prior to entry in this study
* Presence of other comorbid illnesses with an estimated median life expectancy < 5 years
* Evidence of myelodysplasia (MDS); subjects with history of receiving any prior chemotherapy and/or radiotherapy for the treatment of malignant disease, history of greater than 2 months total prior cyclophosphamide for any condition (regardless of dose and route) and/or subjects presenting with abnormal peripheral blood counts require unilateral bone marrow aspiration for pathology, flow cytometry, cytogenetics, and fluorescence in situ hybridization (FISH) MDS panel (per institutional profile) to rule out MDS
* Pregnancy
* Inability to give voluntary informed consent
* Unwilling to use contraceptive methods for at least 15 months after starting treatment
* History of smoking tobacco (or other related/herbal products) in the prior 3 months
* History of prior autologous hematopoietic cell transplantation

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-09-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2024-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leona Holmberg, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (12):
- United States (12):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - University of Colorado, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Boston Medical Center, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - M D Anderson Cancer Center, Houston, Texas
  - The University of Texas Health Science Center, Houston, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

REFERENCES:
- [Derived] Zielonka J, Higuero Sevilla JP. Autologous hematopoietic stem cell transplant for systemic sclerosis associated interstitial lung disease. Curr Opin Rheumatol. 2024 Nov 1;36(6):410-419. doi: 10.1097/BOR.0000000000001050. Epub 2024 Sep 27. PMID 39348419

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (HDIT Autologous PBSCT): STEM CELL MOBILIZATION AND PREPARATION: Patients receive filgrastim SC on mobilization days 1-4 followed by apheresis until a target dose of CD34+ cells >= 2.5 x 10^6/kg are collected. Patients difficult to mobilize with filgrastim alone receive cyclophosphamide IV or *plerixafor SC on mobilization days 1-2 and filgrastim SC on mobilization days 5-7.
  HDIT CONDITIONING: Patients receive high-dose cyclophosphamide IV over 1-2 hours on days -5 to -2 and anti-thymocyte globulin IV on days -5, -3, -1, 1, 3, and 5.
  TRANSPLANTATION: Patients undergo autologous PBSCT on day 0.
  MAINTENANCE THERAPY: Beginning 2-3 months after transplant, patients receive mycophenolate mofetil PO BID for 2 years.
  Anti-Thymocyte Globulin: Given IV
  Autologous Hematopoietic Stem Cell Transplantation: Undergo autologous PBSCT
  Cyclophosphamide: Given IV
  Filgrastim: Given SC
  Laboratory Biomarker Analysis: Correlative studies
  Mycophenolate Mofetil: Given PO
  Peripheral Blood Stem Cell Transplantation: Undergo autologous PBSCT
  Plerixafor: Given SC
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
Period: Overall Study
Arm/Group | Treatment (HDIT Autologous PBSCT)
Started | 21
Completed (one subject withdrew and was not in the analysis) | 20
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: One patient withdrew consent for study while on therapy . So data provided only on 20 patients .
Arm/Group | Treatment (HDIT Autologous PBSCT)
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: EFS of Patients Undergoing Transplant
Description: Event Free Survival (EFS) was defined as survival without meeting the protocol defined endpoint of organ injury (kidney injury requiring renal replacement dialysis for >6 months, sustained LVEF <30%, or sustained decline of FVC >20%).
Time Frame: At 5 years
Population: 20 participants had data collected for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Treatment (HDIT Autologous PBSCT)
Number analyzed (Participants) | 20
participants | 15

2. Secondary Outcome: All-cause Mortality
Description: Defined as any death.
Time Frame: At 5 years
Measure: Number; unit: participants
Arm/Group | Treatment (HDIT Autologous PBSCT)
Number analyzed (Participants) | 20
participants | 3

3. Secondary Outcome: The Number of Participants With Stable or Improved LVEF
Description: By echocardiogram, left ventricle ejection fraction (LVEF) greater than or equal to 30% for greater than or equal to 3 months
Time Frame: From baseline to year 5
Population: 17 participants were able to be assessed for this outcome measure
Measure: Number; unit: participants
Arm/Group | Treatment (HDIT Autologous PBSCT)
Number analyzed (Participants) | 17
participants | 14

4. Secondary Outcome: Number of Participants Requiring Dialysis
Description: Measured by requiring chronic dialysis greater than or equal to 6 months after transplant or required kidney transplant.
Time Frame: From baseline to year 5
Population: 17 participants who were alive post-transplant were assessed for this outcome measure
Measure: Number; unit: participants
Arm/Group | Treatment (HDIT Autologous PBSCT)
Number analyzed (Participants) | 17
participants | 2

5. Secondary Outcome: The Number of Participants With Disease Progression
Description: Chronic renal dysfunction requiring dialysis greater than or equal to 6 months post transplant or requiring kidney transplant, sustained by echo LVEJF <30% for at least 3 months post transplant, or sustained greater than or equal to 3 months decrease of FVC on pulmonary function test (PFT) > 20% post transplant.
Time Frame: baseline to year 5
Population: 17 participants who were alive post-transplant were assessed for this outcome measure
Measure: Number; unit: participants
Arm/Group | Treatment (HDIT Autologous PBSCT)
Number analyzed (Participants) | 17
participants | 5

6. Secondary Outcome: The Number of Participants Who Completed ALL Health Care Utilization as Assessed by UCSD Healthcare Utilization Surveys
Description: UCSD healthcare utilization is a self-report instrument that asks the patient about outpatient and inpatient visits, prescription and non-prescription medications, any surgeries, and major medical expenses during the last 3 months.
Time Frame: From baseline to 5 years
Population: Data were not collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (HDIT Autologous PBSCT)
Number analyzed (Participants) | 20
Participants | 0

7. Secondary Outcome: The Median SHAQ Score
Description: Scleroderma Health Assessment Questionnaire (SHAQ) is a self reported questionnaire with 8 domains including the following scales: pain, patient global assessment, vascular digital ulcers, lung involvement, and gastrointestinal involvement. The SHAQ is a quality of life measure. Each question is scored from 0 (defined as without difficulty), to 3 (defined as unable to do). Some domains are visual analog scales that are measured first and then changed to the 0-3 scale. The individual scores are combined and divided by 8. A higher score indicates worse functionality and changes in the SHAQ is measured as medium change from baseline. The reported medium change can range from -3 to 3. A negative medium change indicates a better outcome.
Time Frame: Baseline to year 4
Population: 17 participants who were alive post-transplant were assessed for this outcome measure
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Treatment (HDIT Autologous PBSCT)
Number analyzed (Participants) | 17
score on a scale | -1.1 [-1.6 to -0.6]

8. Secondary Outcome: The Number of Participants With Improvement in Pulmonary Function
Description: Outcome measure was assessed as the number of participants who had greater than or equal to 3 months a > 10% improvement in predicted FVC or a > 15% improvement in DLCO.
Time Frame: From baseline to year 5
Population: All 17 participants who were alive post transplant were assessed for this outcome measure
Measure: Number; unit: participants
Arm/Group | Treatment (HDIT Autologous PBSCT)
Number analyzed (Participants) | 17
participants
  FVC improvement | 8
  DLCO improvement | 7

9. Secondary Outcome: The Number of Participants With Significant Infectious Complications
Description: Infections of grade 3 or above
Time Frame: Mobilization to Day + 100 post transplant
Measure: Number; unit: participants
Arm/Group | Treatment (HDIT Autologous PBSCT)
Number analyzed (Participants) | 20
participants | 6

10. Secondary Outcome: The Number of Participants With Non-progression Mortality
Description: deaths without relapse of disease
Time Frame: Baseline to year 5
Measure: Number; unit: participants
Arm/Group | Treatment (HDIT Autologous PBSCT)
Number analyzed (Participants) | 20
participants | 2

11. Secondary Outcome: The Number of Participants Who Survived
Time Frame: Baseline to year 5
Measure: Number; unit: participants
Arm/Group | Treatment (HDIT Autologous PBSCT)
Number analyzed (Participants) | 20
participants | 17

12. Secondary Outcome: The Number of Participants Who Had Regimen-related Toxicities
Description: Defined as adverse events (AEs) >= Grade 3 and assessed by the investigator as 1 of the following: unrelated, unlikely, or possibly related to treatment; probably related to treatment; definitely related to treatment.
  The number of participants that experienced Grade 3 or higher adverse events is reported.
Time Frame: Baseline to 1 year post-transplant, grade 3 or higher adverse events
Measure: Number; unit: participants
Arm/Group | Treatment (HDIT Autologous PBSCT)
Number analyzed (Participants) | 20
participants | 15

13. Secondary Outcome: The Median Time of Initiation of Disease-modifying Antirheumatic Drugs (DMARDS) for Relapse After Transplant
Description: The time in months from transplant to starting new therapy not MMF maintenance for relapse disease.
Time Frame: Transplant to year 5
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (HDIT Autologous PBSCT)
Number analyzed (Participants) | 20
months | 13 [0 to 60]

14. Secondary Outcome: Median Time to Treatment Failure
Description: Time to treatment failure is defined as death or initiation of disease modifying antirheumatic drug (DMARD).
Time Frame: From transplant (day 0) to death or disease progression to year 5
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (HDIT Autologous PBSCT)
Number analyzed (Participants) | 20
months | 9 [1.2 to 53]

15. Secondary Outcome: The Number of Participants With Treatment-related Mortality
Description: Defined by death occurring at any time after start of mobilization procedure to day +90 after autologous HCT and definitely or probably resulting from treatment given in the study.
Time Frame: Baseline to Day 90
Measure: Number; unit: participants
Arm/Group | Treatment (HDIT Autologous PBSCT)
Number analyzed (Participants) | 20
participants | 2

16. Secondary Outcome: The Number of Participants Who Completed ALL Work Productivity Survey (WPS)
Description: The first question assesses employment status, type of job for the employed (non-manual, manual or mixed manual/non-manual) and the status of those unemployed (homemaker, retired, student, unable to work due to SSc, unable to work due to non-SSc health problems, or other, i.e. volunteer). The next 3 questions apply only to employed patients and assess absenteeism (full days of work missed due to SSc), presenteeism (days with work productivity reduced by greater than or equal to 50%), and how much SSc interfered with work productivity on a scale of 0-10.
Time Frame: Baseline to year 5
Population: data were not collected
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (HDIT Autologous PBSCT)
Number analyzed (Participants) | 20
Participants | 0

ADVERSE EVENTS:
Time Frame: All cause mortality was assessed up to 5 years. Adverse events (AE) were assessed from the start of mobilization through Day +100 post transplant . Adverse events were assessed from Day +101 through day + 365 post transplant.
Description: AEs (CTCAE 3.0, grades 3-5) were assessed per study protocol excluding expected mobilization and transplant related AEs until day +100 . AE s (CTCAE 3.0, grades 4-5 ) were assessed per study protocol after day +100.
Arm/Group | Treatment (HDIT Autologous PBSCT)
All-Cause Mortality (participants affected / at risk) | 3/20
Serious Adverse Events (participants affected / at risk) | 3/20
Other Adverse Events (participants affected / at risk) | 13/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (HDIT Autologous PBSCT) (N=20)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) — AE term from start of mobilization to day +100
Cardiac disorders (Cardiac disorders) | 1 (2) — cardiomyopathy, cardiac arrest. AE term from start of mobilization to day +100
Multi-system organ failure (General disorders) | 1 (1) — Multi-system organ failure. AE term from start of mobilization to day +100
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) — AE term from start of mobilization to day +100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (HDIT Autologous PBSCT) (N=20)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
ulceration (Skin and subcutaneous tissue disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
hematoma (Vascular disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
hypertension (Vascular disorders) | 2 (2) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
hypotension (Vascular disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
pulmonary embolism (Vascular disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (4) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
Acute Kidney Injury (AKI) (Renal and urinary disorders) | 2 (2) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
hematuria (Renal and urinary disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
neoplasm, benign (General disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
stroke (Nervous system disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
ALT increased (Metabolism and nutrition disorders) | 3 (3) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
anorexia (Metabolism and nutrition disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
hypokalemia (Metabolism and nutrition disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
Elevated GGT (Investigations) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
fever (Immune system disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
gastric hemorrhage (Gastrointestinal disorders) | 2 (2) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
ileus (Gastrointestinal disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
ventricular tachycardia (Cardiac disorders) | 2 (3) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
cardiac arrhythmia's (Cardiac disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
cardiomyopathy (Cardiac disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
Cytokine Rlease Syndrome (Immune system disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
Sepsis (General disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
Respiratory Failure (General disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
Cardiomyopathy (General disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
Acute KIdney Injury (General disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
Pneumonia (Infections and infestations) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
atrial fibrillation (Cardiac disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
Alk Phos (Metabolism and nutrition disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
hyperkalemia (Metabolism and nutrition disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
acidosis (Metabolism and nutrition disorders) | 2 (2) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
AST increased (Metabolism and nutrition disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
creatinine increased (Metabolism and nutrition disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
hyponatremia (Metabolism and nutrition disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.
renal artery aneurysm (Vascular disorders) | 1 (1) — AE term from start of mobilization to day +100. No reportable AE's day + 101-365.

LIMITATIONS AND CAVEATS:
Health Care Utilization by UCSD Healthcare Utilization Survey and Work Productivity Survey: data was not collected as outlined in study.

Only grade 3-5 AE assessed from start of mobilization- Day +100 post tx, excluding expected mobilization and transplant related AE's. No expected AE of grade 3-4 were captured per study.

Also, AE were assessed from Day +101- day + 365 post tx (Grade 4-5). Per study, only grade 4 and 5 were captured. No grade 1-3 AE were captured per study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Protocol Part 1 (pages 1-59) (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/00/NCT01413100/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: Protocol Part 2 (pages 59-130) (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/00/NCT01413100/Prot_SAP_001.pdf